CLINICAL TRIAL: NCT00004426
Title: Study of Gonadotropin Releasing Hormone Agonist Test Using Leuprolide Acetate in Patients With Gonadotropin Deficiency
Brief Title: Leuprolide in Determining the Cause of Gonadotropin Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13361; UCCH-FDR001012
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2000-01

CONDITIONS: Hypogonadism
Keywords: endocrine disorders; hypogonadism; rare disease
MeSH Terms: conditions — Hypogonadism; Endocrine System Diseases; Rare Diseases | interventions — Gonadotropin-Releasing Hormone; Leuprolide

INTERVENTIONS:
Drug: gonadotropin releasing hormone
Drug: leuprolide

SUMMARY:
RATIONALE: The body's response to one injection of leuprolide may provide more information than the standard test for gonadotropin deficiency in determining whether the cause of gonadotropin deficiency is related to the hypothalamus or the pituitary gland.

PURPOSE: Randomized double-blinded clinical trial to study the effectiveness of leuprolide in determining the cause of gonadotropin deficiency.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double blind study. Patients are randomized to receive leuprolide acetate or gonadotropin releasing hormone (GnRH) first, then cross over to receive the other test.

Patients receive one subcutaneous injection of leuprolide acetate or GnRH, then have blood samples drawn periodically. One month later, patients receive the other test.

Another cohort of patients are randomized to receive leuprolide acetate once daily on days 0, 4, and 8, or days 0, 5, and 10.

Patients are followed for up to 2 years.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Prepubertal children with constitutionally delayed puberty At least 2 years retardation of bone age Spontaneously progress into puberty within 1 year Boys: Testes long diameter 2.5-3.5 cm and plasma testosterone 40-300 ng/dL Girls: Breast development, but premenarcheal OR Hypogonadotropinism Delayed onset of pubertal milestones associated with anterior panhypopituitarism OR Kallman's syndrome No spontaneous progression into puberty within 2 years after 6 months replacement sex steroid treatment

--Prior/Concurrent Therapy--

* At least 2 months since prior sex hormone treatment

--Patient Characteristics--

* Age: 14-18 for children with hypogonadotropinism 9-13 for normal children
* Other: No chronic systemic disease No metabolic disease No endocrine disease No growth hormone deficiency

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 1994-08; Study Completion 1998-09

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. Rosenfield, Study Chair — University of Chicago
Locations (1):
- University of Chicago Children's Hospital, Chicago, Illinois, United States